CLINICAL TRIAL: NCT04713631
Title: Phase 2a Randomised Double-blind Placebo-controlled Trial to Assess Safety, Efficacy of Artesunate & Curcumin in Crohn's Disease Patients, Who Continue to Have Mild to Moderate Disease Activity on an Adequate Dose of Azathioprine
Brief Title: Safety and Efficacy of Artesunate & Curcumin in Crohn's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Collaborators: St George's University of London, London, UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-37-EMP-114
Record Dates: First submitted 2020-12-03; First posted 2021-01-19 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease Activity Index (CDAI); Artesunate; Curcumin; Azathioprine
MeSH Terms: conditions — Crohn Disease | interventions — Artesunate; Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Artesunate and Curcumin (Active Comparator): Artesunate 200 mg PO once a day x 2 weeks. Curcumin 2 gm PO once a day x 13 weeks.
  Interventions: Drug: Artesunate; Drug: Curcumin
- Artesunate and Placebo C (Active Comparator): Artesunate 200 mg PO once a day x 2 weeks. Placebo C x 13 weeks.
  Interventions: Drug: Artesunate; Drug: Placebo C
- Curcumin and Placebo A (Active Comparator): Placebo A x 2 weeks. Curcumin 2 gm PO once a day x 13 weeks.
  Interventions: Drug: Curcumin; Drug: Placebo A
- Placebo A and Placebo C (Placebo Comparator): Placebo A x 2 weeks. Placebo C x 13 weeks.
  Interventions: Drug: Placebo A; Drug: Placebo C

INTERVENTIONS:
Drug: Artesunate — Artesunate is approved for the treatment of malaria and is on the World Health Organization list of Essential Medicines. Artesunate has a hemisuccinate group which confers substantial water-solubility and high oral bioavailability and therefore a convenient oral route of administration. Artesunate has a good safety and tolerability profile, having been used to treat millions of adults and children globally.
  Arms: Artesunate and Curcumin; Artesunate and Placebo C
Drug: Curcumin — Curcumin has been used in Indian cuisine and traditional medicine for centuries. It has low solubility in aqueous solution and yields low serum levels following oral administration. In the setting of inflammatory bowel disease where the required site of action is the bowel, systemic absorption may be less relevant. Curcumin and its reduced metabolites undergo conjugation in the liver. Curcumin has a half life of 6-7 hours. It has been found to be safe at oral doses of 2 gm and 3 gm a day in patients with ulcerative colitis, for up to 1 year. In a dose titration study conducted in children with inflammatory bowel disease 2 gm twice daily of curcumin was well tolerated
  Arms: Artesunate and Curcumin; Curcumin and Placebo A
Drug: Placebo A — Artesunate looking placebo
  Arms: Curcumin and Placebo A; Placebo A and Placebo C
Drug: Placebo C — Curcumin looking placebo
  Arms: Artesunate and Placebo C; Placebo A and Placebo C

SUMMARY:
This is a single center phase 2a, randomised double-blind, placebo-controlled factorial design, proof of concept trial. Patients with Crohn's disease who are on an adequate dose of azathioprine and still continue to active disease (CDAI > 150 and c-reactive protein > 6) will be enrolled. Forty patients will be randomised in a 1:1:1:1 ratio into 4 groups in a 2x2 factorial design to receive artesunate 200 mg PO daily for 2 weeks and / or Curcumin 2 gm PO daily for 3 months or placebo. Treatment Curcumin x 13 weeks Placebo C x 13 weeks Artesunate x 2 weeks Group 1 Group 2 Placebo A x 2 weeks Group 3 Group 4 During the treatment period and follow up period patients will be continued on their regular dose of azathioprine and 5-aminosalicylic acid with no change allowed during the study period. Patients will maintain a daily diary of symptoms and adverse events. Scheduled hospital visits with blood and stool tests will be at baseline, week 1, month 1, month 3 and month 6. Primary endpoint will be remission (defined as CDAI < 150) at 3 months

DETAILED DESCRIPTION:
Primary objective: To study the safety, tolerability and efficacy of Artesunate and Curcumin in patients with Crohn's disease, who have ongoing clinical and biochemical evidence of disease activity despite treatment with azathioprine.

Secondary objectives:

1. To investigate the effect of artesunate and curcumin on azathioprine metabolites
2. To investigate the mechanistic pathways through which artesunate and curcumin act

End points:

Primary endpoints

1. Remission of disease as defined by a Crohn's Disease Activity Index (CDAI < 150) at 3 months.
2. Adverse events Secondary end points

<!-- -->

1. Remission (CDAI < 150) after 1 week, 1 month and 6 months
2. Remission or response (reduction in CDAI of >100) after 1 week, 1 month, 3 months and 6 months
3. Change in CDAI score after 1 week, 1 month, 3 months and 6 months
4. Time to remission by patient symptom diary, Harvey Bradshaw score < 5
5. Number of days when the Harvey-Bradshaw index score was less than 5 after 1 week, 1 month, 3 months and 6 months.
6. Change in c-reactive protein and fecal calprotectin after 1 week, 1 month, 3 months and six months
7. Change from baseline, in levels of thiopurine metabolites 6-Thioguanine and 6-methylmercaptopurine after 1 week Exploratory endpoints

1. Change from baseline of tumor necrosis factor-alpha, oxidative stress markers after 1 week, 1 month, 3 months and 6 months DISEASE CONDITION: Crohn's disease in a chronic inflammatory disease of the intestine that is treated with lifelong immunosuppressive medication. After an initial course of steroids to induce control of the disease, maintenance of remission is achieved through long term use of azathioprine. The long term efficacy of azathioprine for maintenance of remission is around 45%.

Need for Alternative Drugs: In the western countries anti-tumor necrosis factor (infliximab and adalimumab) therapy is increasingly being used for disease that does not respond to azathioprine.

Such treatment is very expensive (2.7 lakhs Indian rupee per year for an adalimumab biomimic) and has the potential to reactivate latent tuberculosis (~10%).

POSSIBLE SOLUTION: Recently, several workers have turned their attention to the powerful anti-inflammatory properties of naturally occuring substances such as artemisinins and curcumin. They both have shown promising anti-inflammatory properties in small numbers of patients as well as in animal models. Artesunate has been shown to suppress tumor necrosis factor-α expression and T-helper (Th)1/Th17 responses in a trinitrobenzene sulfonic acid colitis model. Curcumin too, has been shown to have a protective effect in a murine model of dextran sulfate sodium induced colitis, through modulation of tumor necrosis factor-alpha release. It has been studied in patients with active and quiescent ulcerative colitis, and shown to be beneficial when compared to placebo.

Safety data:

ARTESUNATE:

Artesunate is approved for the treatment of malaria and is on the World Health Organization list of Essential Medicines. Artesunate has a hemisuccinate group which confers substantial water-solubility and high oral bioavailability and therefore a convenient oral route of administration. Artesunate has a good safety and tolerability profile, having been used to treat millions of adults and children globally. It has a renal mode of excretion and is rapidly eliminated with a half life of 0.5 to 1.5 hours. The recommended treatment of severe malaria is intravenous artesunate 2.4 mg/kg/dose stat, followed by 2.4 mg/kg/dose at 12 hours, 24 hours and 48 hours. This is followed by an oral regime containing artesunate 200 mg a day (for body wt > 36 kg) for 3 days. Artesunate has been used orally at a dose of 200 mg a day as a neoadjuvant therapy in colorectal cancer for a duration of 2 weeks7

. Artesunate has been used as a daily oral dose of 100 mg for a duration of 1 month in a 12 yr old child with Cytomegalovirus infection. Artesunate has been administered as a daily intravenous dose, initiated at 180 mg and escalated to 240 mg, in a post renal transplant patient for 20 days. Hemolysis may occur 1 to 3 weeks after artesunate administration, and is thought to be caused due to synchronous clearance of once infected erythrocytes. This problem is not anticipated in our study population. Hypersensitivity reactions have been described with oral artesunate (frequency not defined). QT prolongation has been reported with other artemisinin derivatives.

CURCUMIN:

Curcumin has been used in Indian cuisine and traditional medicine for centuries. It has low solubility in aqueous solution and yields low serum levels following oral administration. In the setting of inflammatory bowel disease where the required site of action is the bowel, systemic absorption may be less relevant. Curcumin and its reduced metabolites undergo conjugation in the liver. Curcumin has a half life of 6-7 hours. It has been found to be safe at oral doses of 2 gm and 3 gm a day in patients with ulcerative colitis, for up to 1 year. In a dose titration study conducted in children with inflammatory bowel disease 2 gm twice daily of curcumin was well tolerated.

Dosing plan:

Artesunate 4 mg/kg/dose to a maximum of 200 mg PO daily x 2 weeks. If the patient is less than 50 kg, the dose will be reduced to 150 or 100 mg, ensuring that it does not exceed 4 mg/kg/dose. Curcumin will be started concommitantly at a dose of 2 gm daily and continued for 13 weeks.

INSTRUMENTS TO MEASURE DISEASE ACTIVITY:

Several disease activity indices aimed at measuring severity of disease have been developed. We will use Crohn's DIsease Activity index (CDAI) and Harvey Bradshaw index (HBI) to assess the severity of disease in our study population. The CDAI score which needs a hospital visit will be recorded during each patient visit. The HBI can be calculated from the patient's daily symptom diary which the patients will maintain at home. Patients who discontinue study drugs will also be asked to maintain the symptom diary

Crohn's Disease Activity Index:

CDAI is a disease specific index which considers the activity of Crohns disease in 8 domains, each of which evaluates a specific aspect of CD. The overall score, which ranges from 0 to 600 is the sum of weighted scores of each item, and provides a numerical value of disease activity. It has been in use for over 30 years in clinical trials.

All the parameters used in CDAI are recognized clinical features of CD and were selected by an expert group of Gastroenterologists and as such can be considered to possess content validity. In the majority of circumstances, CDAI reflects disease severity and so can be considered to have content validity. CDAI rise has been noted before exacerbations. It can be considered to possess criterion validity as there is no gold standard to measure against and over the years has become the gold standard in itself.

CDAI has limitations in the paediatric population, patients with stoma and those with strictures.

Components of Crohn's Disease Activity Index (CDAI) 1. No of liquid/soft stools (each day for 7 days) x2 2. Abdominal pain, sum of 7 daily ratings (0 none, 1 mild, 2 moderate, 3 severe) X5 3. General well-being, sum of 7 daily ratings (0 generally well, 1 slightly under par, 2 poor, 3 very poor, 4 terrible) x7 4. Number of listed complications (arthritis or arthralgia, iritis or uveitis, erythema nodosum or pyoderma gangrenosum or aphthous stomatitis, anal fissure or fistula or abscess, other fistula, fever over 37.8°C/100°F) x20 5. Use of diphenoxylate or loperamide for diarrhoea (0 no, 1 yes) X30 6. Abdominal mass (0 no, 2 questionable, 5 definite) X10 7. Haematocrit X6 8. Body weight (1-wt/std wt) [times]100 (add or subtract according to sign) X1 Total score The index score is calculated by adding all the scores. A score <150 is considered as inactive disease; 150-219 mild disease, 220-450 moderately active disease, whilst >450 is considered severe disease. An increase of over 100 from baseline will be considered as relapse for this study. Harvey Bradshaw index (HBI) / modified CDAI The CDAI requires a patient to maintain a 7 day diary which can prove difficult. Mayo Clinic Disease Activity Index looks only at symptoms and signs over the last 24 hours. It also reduces the original 8 components to 5; removing anti-diarrhoeal use, hematocrit level and body weight. The Mayo Clinic Disease Activity Index had a 93% correlation to CDAI in original prospective study of 112 patients.

1. General well-being (0 = very well, 1 = slightly below average, 2 = poor, 3 = very poor, 4

   = terrible)
2. Abdominal pain (0 = none, 1 = mild, 2 = moderate, 3 = severe
3. Number of liquid stools per day
4. Abdominal mass (0 = none, 1 = dubious, 2 = definite, 3 = tender)
5. Complications (1 point for each) - Arthralgia - Uveitis - Erythema Nodosum - Aphthous Ulcers

   - Pyoderma Gangrenosum

   - Anal Fissure
   * New Fistula
   * Abscess Scoring <5 Remission 5-7 Mild Disease 8-16 Moderate Disease >16 Severe Disease Forty patients will be randomised in a 1:1:1:1 ratio in to 4 groups in a 2x2 factorial design to receive artesunate 200 mg PO daily for 2 weeks and / or Curcumin 2 gm PO daily for 3 months or placebo. During the treatment period and follow up period patients will be continued on their regular dose of azathioprine and 5-aminosalicylic acid with no change allowed during the study period. Patients will maintain a daily diary of symptoms and adverse events. Scheduled hospital visits with blood and stool tests will be at baseline, week 1, month 1, month 3 and month 6.

Data that will be recorded daily in the patient diary at home

1. general well being (very well / slightly below par / poor / very poor / terrible)
2. number of loose (liquid or soft) stools a day
3. abdominal pain (none / mild / moderate / severe)
4. abdominal mass
5. extraintestinal manifestations (arthralgia / uveitis / erythema nodosum / aphthous ulcers / pyoderma gangrenosum / active anal fissure / new fistula / abscess)
6. adverse events a. allergic drug reaction b. worsening of the disease more than that expected in the natural disease course i. Rise in CDAI score of > 100 from baseline or Harvey-Bradshaw index of 3 from baseline after 4 weeks from study commencement ii. New onset or aggravation of extraintestinal manifestations, after 4 weeks from enrollment

ELIGIBILITY:
Inclusion Criteria:

* Men or women with a diagnosis of Crohn's disease who are being treated with an adequate, constant dose of azathioprine for at least 3 months (adequate dose is 1 mg/kg in those with low Thiopurine methyltransferase, 2 mg per kg in those with normal Thiopurine methyltransferase)
* Age 18 to 65 yrs
* Crohn's disease of mild to moderate activity (CDAI 150 to 450) and c-reactive protein > 6
* Hemoglobin >9, white blood cells > 3500, platelets > 1,00,000
* Bilirubin < 3, alanine transaminase < 3x upper limit of normal
* Glomerular filtration rate >45
* Normal electrocardiogram

Exclusion Criteria:

* Pregnancy, women who are planning to get pregnant and those unwilling to use contraception
* Lactation
* Bowel surgery with the past 3 months
* Intra-abdominal abscess
* Ileostomy or colostomy
* Change in dose of 5-aminosalicylic acid in the past 4 weeks
* Use of corticosteroids within the past 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Remission of disease | Baseline to 6 months
  Remission of disease as defined by a Crohn's Disease Activity Index (CDAI < 150). The change in response will be studied by studying the change in CDAI after 1 week, 1 month, 3 months and 6 months

SECONDARY OUTCOMES:
Effect of artesunate and curcumin on azathioprine metabolites | Baseline to 1 week
  Change from baseline, in levels of thiopurine metabolites 6-Thioguanine/6-methylmercaptopurine after 1 week
Change in tumor necrosis factor-alpha | baseline to 6 months
  Change in tumor necrosis factor-alpha after 1 week, 1 month, 3 months and six months
Change in C-reactive protein | baseline to 6 months
  Change in C-reactive protein after 1 week, 1 month, 3 months and six months
Change in fecal calprotectin | baseline to 6 months
  Change in fecal calprotectin after 1 week, 1 month, 3 months and six months

CONTACTS AND LOCATIONS:
Overall Officials: Uday C Ghoshal, Principal Investigator — Medical council of India, Association of Indian Universities
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS), Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No
This study will be conducted in the Department of Gastroenterology in collaboration Prof. Devinder Kumar,GastroIntestinal Surgery at St George's, University of London Kingston upon Thames, United Kingdom and in inter-departmental collaborations with the department of Microbiology having patients with clinical suspicion with Crohn's disease and facility for laboratory works.

REFERENCES:
- [Background] Suskind DL, Wahbeh G, Burpee T, Cohen M, Christie D, Weber W. Tolerability of curcumin in pediatric inflammatory bowel disease: a forced-dose titration study. J Pediatr Gastroenterol Nutr. 2013 Mar;56(3):277-9. doi: 10.1097/MPG.0b013e318276977d. PMID 23059643
- [Background] Hou L, Huang H. Immune suppressive properties of artemisinin family drugs. Pharmacol Ther. 2016 Oct;166:123-7. doi: 10.1016/j.pharmthera.2016.07.002. Epub 2016 Jul 10. PMID 27411673
- [Background] Yang Z, Ding J, Yang C, Gao Y, Li X, Chen X, Peng Y, Fang J, Xiao S. Immunomodulatory and anti-inflammatory properties of artesunate in experimental colitis. Curr Med Chem. 2012;19(26):4541-51. doi: 10.2174/092986712803251575. PMID 22834815